CLINICAL TRIAL: NCT02280889
Title: Quality of Life and Experience of Stigmatization in Children with Congenital Melanocytic Nevi Before and After Nevus Excision: a Prospective Study
Brief Title: Quality of Life and Stigmatization in Children with Congenital Melanocytic Nevi Before and After Nevus Excision
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0242; PB_2019-00139 (Other: EC Zurich)
Record Dates: First submitted 2014-10-13; First posted 2014-11-03 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Quality of Life; Stigmatization
Keywords: quality of life; nevus or scar; stigmatization; scar
MeSH Terms: conditions — Stereotyping; Nevus; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Congenital melanocytic nevi (CMN) are a quite common congenital disorder. Over years, surgical excision was proposed to the patients because transformation into a malignant skin tumor (melanoma) was feared. Recent data proof that the risk for malignancy was overestimated. Nowadays still a lot of patients express their wish for surgical removal out of aesthetic reasons and psychological impacts. Many patients and families experience stigmatization because of the nevus. To proof a medical indication for surgical removal the investigators want to evaluate the quality of life and stigmatization before and after nevus surgery.

DETAILED DESCRIPTION:
All children with CMN that will have their nevus removed in our surgical department will be asked to participate. The investigators will send a package of questionnaires to evaluate quality of life and stigmatization before nevus surgery. One year after surgical therapy is finished (sometimes more then one session is necessary), the scar will be clinically evaluated and also another questionnaire package will be sent to evaluate the same parameters again. All parameters are checked for the patients and the families as well. Therefore self and proxy reports of the parents are asked. Moreover, for the patients this is done with interviews in case they are older than 7 years.

ELIGIBILITY:
Inclusion Criteria:

* patients with a congenital melanocytic nevi of at least 2 cm2 that will be removed surgically
* age between 9 months and 16 years

Exclusion Criteria:

* mental retardation of the child
* insufficient knowledge of the German language of both parents
* severe comorbidities
* previous therapies done for the CMN (dermabrasion, surgery, laser)

Ages: 9 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients with CMN of at least 2 square centimeter (projected adult size) that are scheduled for surgical removal of the CMN at our tertiary center for pediatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change of Quality of Life of affected children before and after surgery | Before surgery, up to 90 days after screening and one year after surgery
  Quality of life with the CMN and in comparison with the scar after nevus excision is measured using validated age-related questionnaires respectively one-to one interviews

SECONDARY OUTCOMES:
Change of experiences of stigmatization before and after surgery | Before surgery, up to 90 days after screening and one year after surgery
  Stigmatization experiences of patients and parents before CMN surgery in comparison with after nevus excision are measured using standardized and validated questionnaires
Satisfaction with the treatment | One year after surgery
  Satisfaction with the treatment is evaluated one year after the last surgical step using open questions with rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Neuhaus, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Division of Pediatric Plastic and reconstructive Surgery, Zurich, Switzerland